CLINICAL TRIAL: NCT04534933
Title: Flow Controlled Ventilation Versus Pressure Controlled Ventilation in Thoracic Surgery With One Lung Ventilation - a Prospective, Randomized Clinical Study
Brief Title: Flow Controlled Ventilation in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1014/2020
Record Dates: First submitted 2020-08-13; First posted 2020-09-01 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2020-02

CONDITIONS: Positive-Pressure Respiration, Intrinsic
Keywords: flow controlled ventilation; pressure controlled ventilation; thoracic surgery; one lung ventilation
MeSH Terms: conditions — Positive-Pressure Respiration, Intrinsic

STUDY DESIGN:
Intervention Model Description: controlled, prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCV (Experimental): Artificial ventilation will be performed with individualized flow-controlled ventilation (Evone, Ventinova Medical B.V., Eindhoven, the Netherlands) during thoracic surgery. Individualization will be established by compliance guided end-expiratory and peak pressure setting during two lung ventilation as well as one lung ventilation, flow setting will be adjusted to secure normocapnia during two lung ventilation and the targeted paCO2 during one lung ventilation is 40-60 mmHg, provided that pH >7.2. The I:E ratio will be set to 1:1. The FiO2 will be set to achieve normoxia during two lung ventilation, increased to 100% before lung isolation and after 15 minutes of one-lung ventilation again decreased to secure normoxia or mild hyperoxia (target paO2 of 75-120 mmHg). No recruitment maneuver will be performed for re-inflation of the separated lung and after regain of spontaneous breathing tracheal extubation performed in the operating room.
  Interventions: Device: Evone
- PCV (Active Comparator): Artificial ventilation will be performed with pressure-controlled ventilation (Primus, Dräger, Lübeck, Germany) during thoracic surgery. Peak pressure will be set to achieve a tidal volume of 6-8 ml/kg predicted body weight (PBW) at a compliance titrated positive end-expiratory pressure during two lung ventilation and the tidal volume will be reduced to 4-6 ml/kg PBW during one lung ventilation. Respiratory rate will be set to maintain normocapnia during two lung ventilation and a targeted paCO2 level during one lung ventilation of 40-60 mmHg, provided that pH > 7.2. The I:E ratio will be set to 1:1.5 except extension of expiration is necessary in order to avoid air trapping. The FiO2 will be set to achieve normoxia during two lung ventilation, increased to 100% before lung isolation until 15 minutes of one lung ventilation and decreased thereafter to achieve a targeted paO2 level of 75-120 mmHg. For re-inflation a manual recruitment maneuver will be performed under surgical guidance.
  Interventions: Device: Primus

INTERVENTIONS:
Device: Evone — Airway ventilation device
  Arms: FCV
Device: Primus — Airway ventilation device
  Arms: PCV

SUMMARY:
This trial investigates effects of individualized (by compliance guided pressure settings) flow-controlled ventilation compared to best clinical practice pressure-controlled ventilation in thoracic surgery requiring one lung ventilation.

DETAILED DESCRIPTION:
Flow-controlled ventilation (FCV) is a novel ventilation method with promising first results in porcine studies as well as clinical cross-over trials. A more efficient and maybe lung protective ventilation strategy would be crucial in the challenging situation of one lung ventilation during thoracic surgery, when the whole gas exchange has to be provided by just one half of the lungs.

Thus, individualized FCV, based on compliance guided pressure settings, will be compared to standard of pressure-controlled ventilation in thoracic surgery requiring one lung ventilation in a randomized controlled trial. Based on previous preclinical trials an improvement of oxygenation by 15% will be expected and in order to transfer the preclinical results to humans oxygenation assessed by paO2 / FiO2 ratio after 30 minutes of one lung ventilation is the main primary outcome parameter of this study. Furthermore, improved recruitment of lung tissue due to controlled expiratory flow in FCV will be anticipated without the need of recruitment maneuvers, which may cause deleterious effects on lung tissue. Accordingly any recruitment maneuvers will be omitted in the FCV group.

The investigators hypothesize that improved gas exchange in terms of improved oxygenation and reduced respiratory minute volume required for CO2-removal will be achieved with FCV compared to PCV. Secondary outcome parameters such as the incidence of postoperative pulmonary complications will be additionally assessed in order to plan future studies with clinically relevant outcome.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 18 years
* Body weight ≥ 40 kg
* Elective thoracic surgery requiring OLV
* ASA I-III
* Written informed consent

Exclusion Criteria:

* Emergency surgery
* Female subjects known to be pregnant
* Known participation in another interventional clinical trial
* high pulmonary risk (ppo FEV1<20ml/kg in male or ppo FEV1<18ml/kg in female)
* Empyema evacuation or signs of pulmonary infection
* High grade CMP (EF<30%)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
paO2 / FiO2 ratio (Horowitz Index) | after 30 minutes of one lung ventilation
  Comparison of oxygenation assessed by arterial partial pressure of oxygen (paO2) / fraction of inspired oxygen (FiO2)

SECONDARY OUTCOMES:
decarboxylation (paCO2) | during two lung ventilation in supine position after anesthesia induction (T1) and change to lateral position (T2), after 15 (T3), 30 (T4) and 60 minutes (T5) of one lung ventilation and after reinflation before tracheal extubation (T6)
  Required respiratory minute volume to achieve a taregeted paCO2 of 35-45 mmHg during two lung ventilation and 40-60 mmHg during one lung ventilation
venous admixture (Qs / Qt) | during two lung ventilation in supine position after anesthesia induction (T1) and change to lateral position (T2), after 15 (T3), 30 (T4) and 60 minutes (T5) of one lung ventilation and after reinflation before tracheal extubation (T6)
  Comparison of calculated venous admixure from arterial and central venous blood gas analysis
respiratory minute volume | during two lung ventilation in supine position after anesthesia induction (T1) and change to lateral position (T2), after 15 (T3), 30 (T4) and 60 minutes (T5) of one lung ventilation and after reinflation before tracheal extubation (T6)
  Comparison of respiratory minute volume
respiratory rate | during two lung ventilation in supine position after anesthesia induction (T1) and change to lateral position (T2), after 15 (T3), 30 (T4) and 60 minutes (T5) of one lung ventilation and after reinflation before tracheal extubation (T6)
  Comparison of respiratory rate
tidal volume | during two lung ventilation in supine position after anesthesia induction (T1) and change to lateral position (T2), after 15 (T3), 30 (T4) and 60 minutes (T5) of one lung ventilation and after reinflation before tracheal extubation (T6)
  Comparison of applied tidal volume
positive end-expiratory pressure | during two lung ventilation in supine position after anesthesia induction (T1) and change to lateral position (T2), after 15 (T3), 30 (T4) and 60 minutes (T5) of one lung ventilation and after reinflation before tracheal extubation (T6)
  Comparison of set positive end-expiratory pressure
peak pressure | during two lung ventilation in supine position after anesthesia induction (T1) and change to lateral position (T2), after 15 (T3), 30 (T4) and 60 minutes (T5) of one lung ventilation and after reinflation before tracheal extubation (T6)
  Comparison of set peak pressure
driving pressure | during two lung ventilation in supine position after anesthesia induction (T1) and change to lateral position (T2), after 15 (T3), 30 (T4) and 60 minutes (T5) of one lung ventilation and after reinflation before tracheal extubation (T6)
  Comparison of resulting driving pressure
respiratory compliance | during two lung ventilation in supine position after anesthesia induction (T1) and change to lateral position (T2), after 15 (T3), 30 (T4) and 60 minutes (T5) of one lung ventilation and after reinflation before tracheal extubation (T6)
  Comparison of measured respiratory compliance
applied mechanical power | during two lung ventilation in supine position after anesthesia induction (T1) and change to lateral position (T2), after 15 (T3), 30 (T4) and 60 minutes (T5) of one lung ventilation and after reinflation before tracheal extubation (T6)
  Comparison of calculated applied mechanical power from the ventilator
respiratory resistance | during two lung ventilation in supine position after anesthesia induction (T1) and change to lateral position (T2), after 15 (T3), 30 (T4) and 60 minutes (T5) of one lung ventilation and after reinflation before tracheal extubation (T6)
  Comparison of measured respiratory resistance
heart rate | during two lung ventilation in supine position after anesthesia induction (T1) and change to lateral position (T2), after 15 (T3), 30 (T4) and 60 minutes (T5) of one lung ventilation and after reinflation before tracheal extubation (T6)
  Comparison of measured heart rate
mean arterial pressure | during two lung ventilation in supine position after anesthesia induction (T1) and change to lateral position (T2), after 15 (T3), 30 (T4) and 60 minutes (T5) of one lung ventilation and after reinflation before tracheal extubation (T6)
  Comparison of measured mean arterial pressure
central venous pressure | during two lung ventilation in supine position after anesthesia induction (T1) and change to lateral position (T2), after 15 (T3), 30 (T4) and 60 minutes (T5) of one lung ventilation and after reinflation before tracheal extubation (T6)
  Comparison of measured central venous pressure
Concentration of plamatic cytokine levels | preoperative before induction of general anesthesia and postoperative at PACU admission and 1 hour thereafter
  Plasmatic cytokine level of IL-6, IL-8, IL-10 and TNF-alpha will be assessed pre- (before induction of general anesthesia) and postoperative (ad PACU admission and 60 minutes therafter).
length of PACU stay | Time from PACU admission to transfer to a general ward in hours
  Duration of the patient at the post-anesthesia care unit (PACU)
length of hospital stay | days from surgery to hospital discharge
  Comparison of length of hospital stay after thoracic surgery
postoperative pulmonary complications (PPC) | until hospital discharge or day 30 of hospital stay
  PPC will be assessd daily until hospital discharge or day 30 of hospital stay from the medical records during the follow-up period. The European Perioperative Clinical Outcome (EPCO) definition will be used to assess the occurrence of PPC.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Martini, MD, Principal Investigator — Medical University Innsbruck, Dept. of Anaesthesiology
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Background] Schmidt J, Wenzel C, Mahn M, Spassov S, Cristina Schmitz H, Borgmann S, Lin Z, Haberstroh J, Meckel S, Eiden S, Wirth S, Buerkle H, Schumann S. Improved lung recruitment and oxygenation during mandatory ventilation with a new expiratory ventilation assistance device: A controlled interventional trial in healthy pigs. Eur J Anaesthesiol. 2018 Oct;35(10):736-744. doi: 10.1097/EJA.0000000000000819. PMID 29734208
- [Background] Weber J, Schmidt J, Straka L, Wirth S, Schumann S. Flow-controlled ventilation improves gas exchange in lung-healthy patients- a randomized interventional cross-over study. Acta Anaesthesiol Scand. 2020 Apr;64(4):481-488. doi: 10.1111/aas.13526. Epub 2019 Dec 30. PMID 31828755
- [Background] Weber J, Straka L, Borgmann S, Schmidt J, Wirth S, Schumann S. Flow-controlled ventilation (FCV) improves regional ventilation in obese patients - a randomized controlled crossover trial. BMC Anesthesiol. 2020 Jan 28;20(1):24. doi: 10.1186/s12871-020-0944-y. PMID 31992213